CLINICAL TRIAL: NCT04770454
Title: A Multicenter, Prospective, Non-interventional Observational Study to Evaluate the Quality of Life and Treatment of Anxiety Symptoms of Buspar® Tab (Buspirone) in Patients With Depression Disorder in Korea
Brief Title: Evaluate the Quality of Life and Treatment of Anxiety Symptoms of Buspirone in Patients With Depression Disorders(BASIS)
Acronym: BASIS
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-BPR-OS-401
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Depressive Disorder, Major; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 20 sites in Korea including the Catholic University of Korea, Yeouido St. Mary's Hospital.

Patients with Depressive disorders taking a selective serotonin reuptake inhibitor (SSRI) antidepressant or Serotonin and norepinephrine reuptake inhibitor (SNRI), who additionally administered Buspar® Tab (Buspirone) to control symptom of anxiety.

Primary objective: To evaluate the efficacy of treating the symptoms of anxiety at 12 weeks from the baseline after the administration of Buspar® Tab (Buspirone) to patients with depression by using the Hamilton Anxiety (HAM-A). Approximately 400 participants (including 10% dropouts) Rating Scale

DETAILED DESCRIPTION:
In this study, necessary data will be collected by history taking and medical record review of patients who are taking an SSRI or SNRI antidepressant in the clinical practice and at the same time being additionally administered Buspar® Tab (Buspirone) for the treatment of symptoms of anxiety.

Encourage outpatients with depression accompanied by symptoms of anxiety visiting medical centers in Korea to participate in this study and obtain voluntary consent from them. Have the patients sign the instruction and informed consent form for the use of personal information and enroll them if they meet the inclusion/exclusion criteria. Collect the following data in the case report form (CRF) during the 12-week follow-up observation period.

The HAM-A, HAM-D, and CGI-S are measured at the baseline and at 4, 8, and 12 weeks. The CGI-I is measured at 4, 8, and 12 weeks, and the SDS and WHO-5 are measured at the baseline and at 12 weeks. The following data regarding all the subjects enrolled in this study are collected in the CRF during the 12-week follow-up observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have voluntarily signed the instruction and consent form for the use of personal information
2. Adults over 19 years of age
3. Patients diagnosed with Depressive disorders according to the DSM-5 criteria
4. Patients with a HAM-A score of 18 or higher on the date of enrollment
5. Patients taking an SSRI or SNRI antidepressant at an effective dose or higher for 4 weeks or longer whose symptoms of anxiety are being additionally treated with Buspar® Tab (Buspirone)
6. Patients with the ability to read and understand self-rated scales

Exclusion Criteria:

1. Patients listed in the contraindication group for Buspar® Tab (Buspirone)
2. Patients administered an azapirone class of anxiolytics including buspirone during the last 4 weeks
3. Patients administered a benzodiazepine class of anxiolytics for the first time or with a dose change during the last 1 weeks
4. Patients administered a psychostimulant or medication for attention deficit hyperactivity disorder (ADHD) during the last 4 weeks
5. Pregnant or lactating women
6. Subjects participating in another clinical trial or taking an investigational product for another clinical trial within 12 weeks after the screening visit (Visit 1)
7. Patients determined by the Investigator to be at risk of suicide, self-harm, or hurting others
8. Other subjects determined to be unsuitable by the Investigator

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Depressive disorders taking a selective serotonin reuptake inhibitor (SSRI) antidepressant or Serotonin and norepinephrine reutake inhibitor(SNRI)antidepressant, who additionally administered Buspar® Tab (Buspirone) to control symptom of anxiety.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) score | at 12 weeks
  change from baseline in HAM-A score at week 12 The scale consists of 14 items designed to assess the severity of a patient's anxiety. Each of the 14 items contains a number of symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe. All of these scores are used to compute an overarching score that indicates a person's anxiety severity.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) score | at 4 and 8 weeks
  change from baseline in HAM-A score at week 4,8
  *The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Hamilton Depression Rating Scale (HAM-D) score | at 4, 8, and 12 weeks
  change from baseline in HAM-D score at week 4,8 and 12
  *The Hamilton Depression Rating Scale (HAM-D) contains 17 items (HDRS17) pertaining to symptoms of depression experienced over the past week. For the HDRS17, a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Clinical Global Impression Scale-Severity(CGI-S) | at 4, 8, and 12 weeks
  change from baseline in CGI-S score at week 4,8 and 12
  *The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Clinical Global Impression Scale-Improvement(CGI-I) | at 4, 8, and 12 weeks
  Score at week 4,8 and 12 point after medication
  *The CGI-Improvement (CGI-I) is similarly simple. Each time the patient is seen after medication has been initiated, the clinician compares the patient's overall clinical condition to the one week period just prior to the initiation of medication use (the so-called baseline visit). Only the following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."
Sheehan Disability Scale(SDS) score | at 12 weeks
  change from baseline in SDS score at week 12
  *Sheehan Disability Scale(SDS) generates 4 scores: a work disability score, a social life disability score, a family life disability score and a total score. To get a total score add up the 3 individual scores (work: social life: family life). The maximum possible score is 30.
5-item World Health Organization Well-Being Index(WHO-5) | at 12 weeks
  change from baseline in WHO-5 score at week 12
  *WHO-5 Well-being Index (WHO-5) consists of five positively worded items that are rated on 6-point Likert scale, ranging from 0 (representing worst possible) to 5 (representing best possible quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- the Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul, Yeouido, South Korea

IPD SHARING:
Plan to Share IPD: No